# GlaxoSmithKline Biologicals SA

## 218595

A Phase 1, Open-label, Safety and Immunogenicity Study of a Booster Dose of the Investigational CV0501 mRNA COVID-19 Vaccine in Adults at Least 18 Years Old 31Jan2023

Statistical Analysis Plan

Version 3.0

Prepared by:

PPD, part of Thermo Fisher Scientific

Granta Park Great Abington CB21 6GQ Cambridge, UK

# VERSION HISTORY

| Version | Date | Details |
|----------|-----------|-----------------------------------------------|
| SAP v1.0 | 12MAY2022 | Prepared for IND submission |
| SAP v2.0 | 19AUG2022 | Updated for protocol amendments 1 (23JUN2022) |
| | | and 2 (26JUL2022) |
| SAP v3.0 | 31JAN2023 | Updated based on changes to ANCOVA model and |
| | | prior Covid-19 infection incorporated into |
| | | immunogenicity and Demography summaries. |



# TABLE OF CONTENTS

| LI | ST OF ABBREVIATIONS | VI |
|---|---|---|
| 1. | INTRODUCTION | 1 |
| 2. | OBJECTIVES | 2 |
| 2.1.<br>2.2.<br>2.3. | PRIMARY OBJECTIVE AND ENDPOINTS | 2 |
| 3. | INVESTIGATIONAL PLAN | 3 |
| 3.1.<br>3.2.<br>3.3.<br>3.4. | OVERALL STUDY DESIGN AND PLAN STUDY ENDPOINTS TREATMENTS Dose Adjustment/Modifications | 6 |
| 4. | GENERAL STATISTICAL CONSIDERATIONS | 7 |
| 4.1.<br>4.2.<br>4.3.<br>4.3.1. | | 8<br>9<br><i>9</i> |
| 4.3.2.<br>4.3.3. | · F | |
| 5. | PARTICIPANT DISPOSITION | 9 |
| 5.1.<br>5.2. | DISPOSITION | 10 |
| 6.1. | DEMOGRAPHICS | |
| 6.2.<br>6.3. | Baseline Disease Characteristics 1 Medical History 1 General Medical History 1 | 11<br>12 |
| 6.4. | INCLUSION AND EXCLUSION CRITERIA | 12 |
| 7. | TREATMENTS AND MEDICATIONS | 12 |
| 7.1.<br>7.1.1.<br>7.1.2.<br>7.2. | | |
| 7.2.1 | | |
| 8. | ANALYSIS OF SAFETY AND IMMUNOGENICITY STUDY OBJECTIVE | S14 |
| findir | ANALYSIS OF PRIMARY SAFETY OBJECTIVE | y 1-7),<br>aboratory<br>ents (Day 1 – |

| 8.2.1. GM/s of neutralizing Ab titer against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 and GM/ from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers = 12 8.3. ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS 15 8.4.1 | 9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.2<br>9.3<br>9.4<br>9.5 | Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
|---|---|---|---|
| Omicron BA 1, BA 2 and BA 5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA 1, BA 2 and BA 5 variants at each collection time point 14 8.22. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA 1, BA 2 and BA 5 variants at each collection timepoint, with seroresponse defined as postboost fiters ≥ 4× preboost fiters. 12 8.3 ANALYSIS OF EXPLORATORY IMMUNOGENICITY ENDPOINTS 15 8.4 ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS 16 8.4.1 Service Adverse Events 17 9 SAFETY ANALYSIS 19 9.1 ADVERSE EVENTS 19 9.1.1 Relationship of Adverse Events to Study Drug 20 9.1.2 Severity or Adverse Event 20 9.1.4 Solicited Adverse Event 22 9.1.4 Solicited Adverse Event 22 9.1.5 Unsolicited Adverse Event 22 9.1.6 Adverse Events 22 9.1.7 Serious Adverse Event 22 9.1.8 Medically Attended Adverse Event 22 9.1.9 Adverse Events Leading to Treatment Discontinuation 24 9.1.1 Death 24 9.2 CLINICAL LABORATORY EVALUATIONS 26 9.3 VITAL SIGN MEASUREMENTS 26 9.4 PHYSICAL EXAMINATION 26 9.5 ELECTROCARDIOGRAM 26 | 9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.2<br>9.3<br>9.4<br>9.5 | Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline or neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as posiboost filters ≥ 4× preboost filters. 12 8.3. ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS. 15 8.4.1 CC 1 17 8.4.2 CC 1 18 9. SAFETY ANALYSIS 19 9.1 ADVERSE EVENTS 19 9.1.1 Relationship or Adverse Events to Study Drug 20 9.1.2 Severity or Adverse Events Los Study Drug 20 9.1.3 Outcome or Adverse Event 22 9.1.4 Solicited Adverse Event 22 9.1.5 Unsolicited Adverse Event 22 9.1.6 Adverse Events or Special Interest 22 9.1.7 Serious Adverse Events Leading to Treatment Discontinuation 22 9.1.8 Medically Attended Adverse Events Leading to Study Discontinuation 22 9.1.1 Death 22 9.2 CLINICAL LABORATORY EVALUATIONS 25 9.3 VITAL SIGN MEASUREMENTS 26 9.4 PHYSICAL EXAMINATION 26 | 9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.2<br>9.3<br>9.4 | Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as posiboost fiters ≥ 4× preboost fiters. 12 8.3. ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS. 15 8.4.1 CC 15 9. SAFETY ANALYSIS 19 9.1 ADVERSE EVENTS 19 9.1.1 Relationship or Adverse Events to Study Drug 20 9.1.2 Severity or Adverse Events | 9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.2<br>9.3<br>9.4 | Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of noutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers. 15 8.3 ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS 15 8.4 ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS 15 8.5 ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS 16 8.4.1 CCI 16 8.4.1 CCI 17 8.4.2 CCI 17 9 SAFETY ANALYSIS 19 9.1 ADVERSE EVENTS 19 9.1.1 Relationship or Adverse Events to Study Drug 20 9.1.2 Severity of Adverse Events 19 9.1.2 Severity of Adverse Event 20 9.1.3 Outcome or Adverse Event 20 9.1.4 Solicited Adverse Event 22 9.1.5 Unsolicited Adverse Event 22 9.1.6 Adverse Events or Special Interest 22 9.1.7 Serious Adverse Events 22 9.1.8 Medically Attended Adverse Events 22 9.1.9 Adverse Events Leading to Treatment Discontinuation 24 9.1.10 Adverse Events Leading to Study Discontinuation 24 9.1.11 Death 22 9.2 CLINCAL LABORATORY EVALUATIONS 25 9.3 VITAL SIGN MEASUREMENTS. 25 | 9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.1.<br>9.2<br>9.3 | .6 Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as posiboost titers ≥ 4× preboost titers. 12 8.3. ANALYSIS OF TERTIARY IMMUNOGENICITY ENDPOINTS. 15 8.4. ANALYSIS OF EXPLORATORY IMMUNOGENICITY ENDPOINTS. 16 8.4.1 CI 8.4.2 CI 9 SAFETY ANALYSIS | 9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 2 | 6 Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers | 9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 1. | 6 Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost fiters ≥ 4× preboost fiters | 9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 1. | .6 Adverse Events of Special Interest | 22<br>23<br>24<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost filters ≥ 4× preboost filters | 9. 1.<br>9. 1.<br>9. 1.<br>9. 1.<br>9. 1. | 6 Adverse Events of Special Interest | 22<br>22<br>23<br>24 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab liters against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.22. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab liters against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost filters | 9. 1.<br>9. 1.<br>9. 1.<br>9. 1. | .6 Adverse Events of Special Interest | 22<br>22<br>23 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers | 9. 1.<br>9. 1. | .6 Adverse Events of Special Interest | 22<br>22 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers | 9.1. | | 22 |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline or neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers | | O DOMESTICA FRANCISCO E VENE INTERNATIONAL I | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers | q 1 | | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers \(\geq 4\times \text{ preboost titers.}\) | | | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers | | | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers $\geq$ 4× preboost titers | | | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers $\geq$ 4× preboost titers | | | _ |
| Omicron BA. 1, BA. 2 and BA. 5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA. 1, BA. 2 and BA. 5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA. 1, BA. 2 and BA. 5 variants at each collection timepoint, with seroresponse defined as postboost titers \geq 4 \times preboost titers | | | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers \geq 4 \times preboost titers | | | 18 |
| Omicron BA. 1, BA. 2 and BA. 5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA. 1, BA. 2 and BA. 5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA. 1, BA. 2 and BA. 5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4 × preboost titers | | | |
| Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point 14 8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers \(\geq 4\times preboost titers | | | |
| 0.2.1. Olvirs of fleditalizing no liter against pseudotyped bearing 5 protein from 5/105 00 v 2 vv i, | poir<br>8.2.<br>psec<br>coll<br>8.3 | vicron BA. 1, BA. 2 and BA. 5 and GMI from baseline of neutralizing Ab titers against pseudotyped oring S protein from SARS-CoV-2 WT, Omicron BA. 1, BA. 2 and BA. 5 variants at each collection int 14 and 14 and 15 and 1 | ime<br>jainst |
| | | . 2. 22 2. 2. 2. 2. 2. 2. Constitution and the study in the study in the | 14 |
| 8.1.2. Analysis of Medically attended Adverse Events (MAAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) from study vaccination through the end of the study | Aav<br>8.2.<br>8.2. | | |

| GlaxoSmithKline Biologicals SA<br>CV2 SARS-CV0501-012 BST (218595) | | |
|---|---|---|
| | 13 | CHANGES IN THI |

| 13 | CHANGES IN THE PLANNED ANALYSIS | |
|---|---|---|
| 14 | REFERENCES | |
| 15 | APPENDICES | |
| 15.2 K | SCHEDULE OF EVENTS<br>KNOWN LLOQS AND ULOQS FOR DIFFERENT ASSAYS<br>MEDDRA QUERIES FOR IDENTIFYING AESIS | 30 |
| Figure 3-1 | LIST OF FIGURES Study Design Part A | 5 |
| | Study Design Part B | |

Statistical Analysis Plan Date Issued: 31JAN2023

# List of Abbreviations

| Abbreviation | Definition |
|---|---|
| AE | adverse event |
| AESI | adverse event of special interest |
| ANCOVA | analysis of covariance |
| BMI | body mass index |
| CI | confidence interval |
| CCI | CCI |
| COVID-19 | coronavirus disease |
| CSR | clinical study report |
| CV0501 | an investigational, monovalent, nucleoside-modified, mRNA COVID-19 vaccine targeting the Omicron variant of SARS-CoV-2 |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eDiary | electronic diary |
| EOS | end of study |
| FtiH | first-time-in human |
| GM | Geometric Mean |
| GMI | geometric mean increase |
| GMT | geometric mean titer |
| ICF | informed consent form |
| ICS | intracellular staining assay |
| IgG | immunoglobulin g |
| IP | investigational product |
| IMP | investigational medicinal product |
| LLOQ | lower limit of quantification |
| LNP | Lipid nanoparticles |
| MAAE | medically attended adverse event |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mRNA | messenger ribonucleic acid |
| NA | not applicable |
| NAb | Neutralizing antibody |
| N protein | nucleocapsid protein |
| PBMC | peripheral blood mononuclear cell |
| PP | Per protocol |
| PPI | Per protocol Immunogenicity |

| Abbreviation | Definition |
|--------------|-------------------------------------------------|
| PT | Preferred Term |
| SAP | statistical analysis plan |
| RT-PCR | reverse transcription polymerase chain reaction |
| S protein | spike protein |
| SAE | serious adverse event |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SOC | system organ class |
| SRT | Safety Review Team |
| TLF | Table, Listing and figures |
| Th | T helper |
| ULOQ | Upper limit of quantification |
| WHO | World Health Organization |
| WT | Wild type |

#### 1. Introduction

The COVID-19 pandemic caused by SARS-CoV-2 virus was declared by the WHO on 11 Mar 2020 (WHO 2020). As of 19 Jan 2022, more than 332 million cases have been reported worldwide, leading to more than 5.5 million deaths (WHO 2022). To date, there are multiple licensed or conditionally approved vaccines available that rely on a variety of vaccine technologies. All currently available vaccines are based on antigens from the original Wuhan strain (D614; wild-type, hereafter referred to as "WT").

This is a Phase 1 FTiH study designed to evaluate the safety, reactogenicity, and immunogenicity of the GSK-CureVac CV0501 modified mRNA vaccine encoding the Omicron variant to prevent COVID-19. This study will evaluate the CV0501 vaccine as a booster vaccination in a healthy adult population of participants who have previously received at least 2 doses of an mRNA COVID-19 vaccine.

GSK and CureVac are collaborating to develop CV0501, a modified-nucleotide mRNA vaccine based on the same LNP. platform as the CVnCoV vaccine. The CV0501 mRNA encodes S protein from the Omicron variant and has been optimized to improve intracellular mRNA stability and translation for increased and extended protein expression, relative to unmodified S protein mRNA

This statistical analysis plan (SAP) was developed to provide the details of the planned statistical methodology for the analysis of both interim analyses and the preparation of the final clinical study report (CSR).

This SAP is based upon the following study documents:

- Study Protocol CV2 SARS-CV0501-012 BST (218595) Protocol Amendment 2 (26 Jul 2022)
- Participant Case Report Form (25 Jan 2023)

This SAP is to be finalized prior to first participant first visit. Major changes in the analysis that are made after database lock will be documented in the CSR along with the rationale and other details regarding the changes.

# 2. Objectives

# 2.1. Primary Objective and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary – Safety | |
| To evaluate the safety and tolerability of CV0501 at each dose level | Percentage of participants with each solicited local and systemic AEs during 7 days after vaccination (i.e., the day of study vaccination and 6 subsequent days (day 1 through 7) |
| | Percentage of participants with each abnormal clinical<br>safety laboratory finding for 8 days after study<br>vaccination |
| | <ul> <li>Percentage of participants with unsolicited AEs for 28<br/>days after study vaccination</li> </ul> |
| | <ul> <li>Percentage of participants with MAAEs, AESIs and<br/>SAEs from study vaccination through the end of the<br/>study (for 180 days after the study vaccine<br/>administration), each summarized separately</li> </ul> |

# 2.2. Secondary Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Secondary – Immunogenicity | |
| To evaluate neutralizing Ab titers against SARS-CoV-2 WT, Omicron, and Delta* variants following CV0501 booster vaccination in adult participants | <ul> <li>GMTs of neutralizing Ab titers against pseudovirus bearing S protein from SARS-CoV-2 WT, Omicron, and Delta variants at each collection timepoint</li> <li>GMI from baseline of neutralizing Ab titers against pseudovirus bearing S protein from SARS-CoV-2 WT, Omicron, and Delta variants at each collection time point</li> </ul> |
| To describe seroresponse to CV0501 based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron, and Delta* variants | Seroresponse rate 28 days after the booster dose (day 29) based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron, and Delta variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers |

Statistical Analysis Plan Date Issued: 31JAN2023



## 3. Investigational Plan

## 3.1. Overall Study Design and Plan

This open-label, dose escalation first-time-in human (FtiH) Phase 1 study will evaluate the safety (including reactogenicity) and immunogenicity of a single booster dose of CV0501 vaccine in adults who have previously received at least 2 doses of an mRNA COVID-19 vaccine. Approximately 180 participants will be enrolled. The study will comprise two parts (Part A and Part B).

Part A: Participants in Cohorts 1 to 5 will be enrolled in a staggered manner to 1 of 5 cohorts with planned dose escalation of CV0501 from 12  $\mu$ g up to 200  $\mu$ g. Each cohort of Part A will evaluate a single dose level of CV0501 vaccine and will include 2 age groups (younger adults,  $\geq$  18 to < 65 years old, and older adults,  $\geq$  65 years old), as indicated in Table 3-1. The dose levels for the groups in Cohorts 1-3 are fixed. The dose levels for the Cohorts 4 and 5 will be as recommended by the SRT, based on their review of all available safety data and dosing scenarios.

Part B: Designed to comprise 2 single age group cohorts (≥18 to <65 years old), will start based on the first interim analysis of safety and immunogenicity, provided that the SRT assesses the 12µg dose to be immunogenic and safe. The SRT may recommend dropping Cohorts 6 and 7 (Groups 6a and 7a) based on immunogenicity data from the groups that received the 12µg dose level. If the SRT determines that enrollment in Cohorts 6 and 7 may proceed, enrollment may proceed in parallel according to Table 3-2.

Table 3 1 Study Cohorts, Groups, and Study Vaccine Administration (Part A)

| Cohor<br>t | Vaccin<br>e | Dose Level | Group A<br>Younger Adults<br>≥18 to <65 Years of<br>Age<br>(n range) | Group B<br>Older Adults<br>≥65 Years of Age<br>(n range) | Total Cohort<br>Sample Size |
|---|---|---|---|---|---|
| 1 | | 12 μg | 1a (min 10; max 20) | 1b (min 10; max 20) | 30 |
| 2 | | 25 μg | 2a (min 10; max 20) | 2b (min 10; max 20) | 30 |
| 3 | CV050 | 50 μg | 3a (min 10; max 20) | 3b (min 10; max 20) | 30 |
| 4 | 1 | 75 or 100* μg | 4a (min 10; max 20) | 4b (min 10; max 20) | 30 |
| 5 | | 100,150, or 200*<br>μg | 5a (min 10; max 20) | 5b (min 10; max 20) | 30 |

<sup>\*</sup>Depending on the reactogenicity/safety findings from groups in Cohorts 1-3, the SRT may recommend 1 of 3 prespecified dosing scenarios comprising these dose levels for groups in Cohorts 4 and 5, as described in Section 3.1.1 of protocol. The dose level recommendations will be made independently for Groups A (younger participants) and B (older participants).

Table 3 2 Study Cohorts, Groups, and Study Vaccine Administration (Part B)

| Cohor<br>t | Vaccine | Dose<br>Level | Group A Younger Adults ≥18 to <65 Years of Age (n range) | Total Cohort Sample<br>Size |
|---|---|---|---|---|
| 6 | CV0501 | 3 μg | 6a | 15 |
| 7 | CV0501 | 6 μg | 7a | 15 |

Figure 3-1 Study Design Part A



Figure 3-2 Study Design Part B



## 3.2. Study Endpoints

Please refer to Section 2.1 of this SAP.

#### 3.3. Treatments

Investigational product (IP) in this Phase 1 study refers to the CV0501 vaccine, which is a formulation of modified mRNA encoding Omicron variant S protein microencapsulated in lipid nanoparticles (LNP) that will be administered during the study.

The LNPs are composed of a

The following IP will be used in the study:

| Intervention Name | CV0501 |
|---|---|
| Туре | Vaccine |
| Dose Formulation | Modified mRNA |
| Unit Dose Strength(s) | CCI μg mRNA/mL |
| Dosage Level(s) | 3, 6, 12, 25, 50, 75, 100, 150, 200 μg |
| Route of Administration | Intramuscular injection |
| Diluent | 0.9% sodium chloride |
| Use | Experimental |
| IMP or NIMP | IMP |
| Sourcing | Provided centrally by GSK Biologicals SA or CureVac GmbH |
| Packaging and Labeling | IP will be provided in a glass vial as a sterile colloidal |
| | dispersion in a frozen liquid formulation as open-label supply. |
| | Each vial will be labeled as required per country requirement. |

Statistical Analysis Plan Date Issued: 31JAN2023

## 3.4. Dose Adjustment/Modifications

An overdose is any dose of study vaccine given to a participant that exceeds the planned dose for an individual within a given dose group.

There is no specific treatment recommended for an overdose. Overdose itself is not to be reported as an adverse event (AE). Overdose participants will be included in the Safety Set and excluded from Per protocol Immunogenicity (PPI) Set.

## 4. General Statistical Considerations

Participants will be identified in the listings by the participant identification number concatenated with the site number. Data will be displayed in all listings sorted by age group, dose group and participant number.

**Continuous data** will be described using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum).

Categorical data will be described using the participant count and percentage for each category.

For the **summary statistics** of all numerical variables unless otherwise specified, mean, confidence interval, median, standard deviation, minimum and maximum will be displayed.

A row denoted "Missing" will be included in count tabulations where specified on the shells to account for dropouts and missing values.

There is no formal hypothesis testing in this study where statistical methods are applied, the emphasis will be on estimation with 2-sided 95% Confidence intervals (CIs).

The denominator for all percentages will be the number of participants with non-missing values of corresponding parameter in that treatment within the analysis population of interest, unless otherwise specified.

A table, figure, listing (TLF) is to be generated for any required item even where no data is available or reported. In such cases, the table, figure or listing will state: "**No Data Reported**". This will confirm to the health authorities that all data for the tables, figures, listings, and narratives are accounted for.

**Baseline** will be defined as the last non-missing evaluation prior to study vaccine administration, unless otherwise specified.

Study day will be calculated as follows:

- study day prior to the injection will be calculated as: date of assessment date of the injection
- study day on or after the date of the injection will be calculated as: date of assessment date of the injection + 1

For Safety assessment of AEs, the intervals will be calculated as follow

Statistical Analysis Plan Date Issued: 31JAN2023

- solicited AEs: the day of vaccination and 6 subsequent days (day 1 through 7)
- unsolicited AEs: the day of vaccination and 28 subsequent days (day 1 through 28)
- Medically attended adverse events (MAAEs), adverse events of special interest (AESI) and serious adverse events (SAEs): the day of vaccination and 180 subsequent days (day 1 through 180)

For calculations regarding antibody levels/titers, antibody results released as below a value will be replaced by  $0.5 \times$  the value. Results released as above a value will be converted to the value. Missing results will not be imputed.

The lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) for WT NAb are the following:

LLOQ = To be defined by lab when assay calibrated.

ULOQ = To be defined by lab when assay calibrated.

calibrating conversion factor to WHO standard is 1/1.872.

NAb Result (IU/mL) = Result (NT50 titer) x 1/1.872.

Details on LLOQs and ULOQs for IgG and conversion factors when available are described in Section 15.2 All safety data summaries/displays will be provided by dose group. Details will be included in the TLF shell. All statistical analyses will be performed using SAS® software Version 9.4 or later.

## 4.1. Sample Size

The sample size is based on clinical considerations to inform dose regimen decisions for continued clinical development.

Approximately 180 participants will be enrolled in this Phase 1 study, 5 dose-level cohorts (Cohorts 1 to 5) each comprising 2 age groups. Cohorts 6 and 7 will comprise 1 age group (younger adults). With 30 participants in each cohort, there is a 78.5% probability to observe at least 1 AE if the incidence rate is 5% and a 95.8% probability to observe at least 1 AE if the incidence rate is 10%. With 30 participants in each cohort, a 10% unevaluable rate for immunogenicity results, and a standard deviation of 0.45 for log10-transformed increase from day 1, the ratio of the upper limit of a 2-sided 95% CI and the point estimate of geometric mean increase (GMI) is 1.5. The sample size in Cohorts 6 and 7 is based on clinical feasibility rather than on statistical rationale. With 15 participants in each cohort, there is a 79.4% probability to observe at least one AE if the true incidence rate is 10%.

## 4.2. Randomization, Stratification, and Blinding

Participants in Part A will be assigned sequentially to a dose-level cohort by age group. Participants in Part B will be randomly assigned on day 1 to receive study vaccine by dose-level cohort.

The study will be open label.

#### 4.3. Analysis Set

The following analysis sets have been defined: Enrolled Set, Per protocol Immunogenicity Set, and Safety Set.

#### 4.3.1. Enrolled Set

The Enrolled Set will include all eligible participants who gave informed consent, regardless of the participants' treatment status in the study.

## 4.3.2. Per protocol Immunogenicity (PPI) Set

The PPI Set includes all eligible participants who received a dose of study IP per protocol and who have values for predose and Day 15 neutralizing Ab titers against pseudovirus bearing S protein from the Omicron BA1 variant of SARS-CoV-2. Results from a blood sample deviating from the dosing or blood sampling schedule and results from a blood sample after intercurrent conditions that may interfere with immunogenicity (e.g., laboratory-confirmed SARS-CoV-2 infections or immunosuppressive or immunodeficient conditions) or after a prohibited concomitant medication/vaccination (COVID-19 vaccination) will be excluded from the PPI Set. The data will be analyzed according to the dose that participants received at Visit 1.

The PPI Set will be used for the immunogenicity analyses.

## 4.3.3. Safety Set

All participants who receive 1 dose of IP. The Safety Set will be used for all analyses of safety. Data are analyzed according to treatment received.

## 5. Participant Disposition

#### 5.1. Disposition

Participant disposition will be summarized by dose group for all participants. The number and percentage of participants for the following categories will be presented: participants who were enrolled, vaccinated, participants who discontinued from the study (i.e. did not complete the day 181 visit), participants in the Enrolled Set, PPI Set and Safety Set.

A participant may withdraw or be withdrawn from the study for any of the following reasons:

- Participant request.
- Investigator request.
- The participant is noncompliant with the protocol.
- The participant has a serious or intolerable AE(s) that, in the investigator's opinion, requires withdrawal from the study.
- The participant is lost to follow-up.

Statistical Analysis Plan Date Issued: 31JAN2023

- Death.
- The sponsor terminates the study.
- The participant has safety laboratory results that reveal clinically significant hematological or biochemical changes from the baseline values, per investigator judgment
- The participant has symptoms or an intercurrent illness not consistent with the protocol requirements or that justify withdrawal
- Other reasons (e.g., pregnancy, development of contraindications of use of the IP)
- The participant withdraws consent, or the investigator or sponsor decides to discontinue their participation in the study withdrawal of consent by participant or the investigator or sponsor decides to discontinue their participation in the study

Participant status summary will also be provided which include participants who completed each visit, participants vaccinated with study vaccine, participants who had immunogenicity results at applicable visit, and participants who completed the study. Participant status summary will be also presented by dose and age group.

Participant disposition and discontinuation data will be presented in a listing sorted by age, dose group and participant number.

The number of participants included in each analysis set will be summarized. A listing of participants in each analysis set will also be provided by age, dose group and participant number. Participants excluded from the analysis sets will be listed with reason for exclusion(s) and sorted by age, dose group and participant number.

The primary reason for study discontinuation includes: Withdrawal due to AE, Lost To Follow-up, Physician Decision, Pregnancy, Site Terminated by Sponsor, Study Terminated by Sponsor, Withdrawal of Consent by Participant, Protocol Deviation, Vaccine Not Administered, Death, Other.

#### **5.2. Protocol Deviations**

Major protocol deviations are a subset of protocol deviations that may significantly impact the completeness, accuracy, or reliability of the study data or that may significantly affect a participant's rights, safety, or well-being. Major protocol deviations rules will be developed and finalized before database lock.

Major protocol deviations include, but are not limited to, the following:

- Study vaccine not administered at all
- Invalid/missing informed consent
- Fraudulent data
- Administration of concomitant vaccine(s) forbidden in the protocol
- Participants got vaccinated but not as per protocol

Statistical Analysis Plan Date Issued: 31JAN2023

- Vaccine storage temperature deviation which is not accepted by quality
- Expired vaccine administered
- Ineligible participant
- Administration of any medication forbidden by the protocol
- Participants did not comply with blood sample schedule
- Serological results not available pre and post-vaccination (day 15 and day 29) for neutralizing Abs against pseudovirus bearing S protein from Omicron BA.1 SARS-CoV-2
- Serological results available but results unreliable (e.g. wrong blood sample management)
- Intercurrent condition impacting immunogenicity

The number of participants with major protocol deviations will be summarized by dose group. Major protocol deviations will be listed with date of occurrence, deviation description, and analysis set from which participant is excluded. Major protocol deviation summary will be based on the Enrolled Set.

The major protocol deviations will be listed by age group, dose group, participant number and reported in the CSR.

## 6. Demographics and Baseline Characteristics

## 6.1. Demographics

A summary of demographics and baseline information will be presented by dose group in each age group. The demographic characteristics consist of age (years), gender at birth, ethnicity, and race. The baseline characteristics consist of height (cm), weight (kg), BMI (kg/m²), N protein, and prior Covid-19 infection, defined as either self reported Covid-19 infection or a positive N protein result from the last result/test prior to vaccination.

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for age, height, weight, and BMI will be provided by study vaccine in each age group and overall.

The number and percentage of participants will be provided for gender at birth, ethnicity, race, prior Covid-19 infection and baseline N protein status by dose group in each age group and overall.

Percentages will be based on the total number of participants in the analysis set defined in the output.

Participant demographic and baseline characteristics will be sorted by age group, dose group and participant number, including child-bearing potential (applicable only for women).

#### 6.2. Baseline Disease Characteristics

Not applicable

Statistical Analysis Plan Date Issued: 31JAN2023

## **6.3. Medical History**

## 6.3.1. General Medical History

Medical history will be coded using the latest version of Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of participants with any medical history, medical history that ended before Visit 1, and medical history that is still ongoing at Visit 1 (at the time of first vaccination) will be summarized overall and for each system organ class (SOC) and preferred term (PT) by dose group. Percentages will be calculated based on safety set.

Participant medical history data including specific details will be presented in a listing sorted by age group, dose group and participant number.

#### 6.4. Inclusion and Exclusion Criteria

Enrolled participants who failed any inclusion/met any exclusion criteria will be classed as major protocol deviations.

#### 7. Treatments and Medications

#### 7.1. Prior and Concomitant Medications

All medications/vaccination will be coded according to the World Health Organization (WHO) drug dictionary (WHODrug), which will be updated whenever available throughout the study.

#### 7.1.1. Prior Medications

Any medications (including vaccines) that were administered to the participant within 6 months of Screening will be considered as prior medication for this study.

Prior medication will be listed sorted by age group, dose group, participant number and summarized by dose groups using the Safety Set. They will be summarized by the generic preferred name and anatomical therapeutic chemical (ATC) class level 4. More than one ATC class per medication is possible and the medication will be reported under all applicable classes. A participant with multiple occurrences within an ATC is counted only once for that ATC class. Similarly, a participant with multiple occurrences within a generic preferred name is counted only once.

#### 7.1.2. Concomitant Medications

Concomitant medications are defined as any medications and vaccine (other than study vaccines) taken after the study vaccine is administered and:

Statistical Analysis Plan Date Issued: 31JAN2023

- Within 6 months of Screening or
- Were taken first prior to the dosing and on-going after study vaccine dose up to 6 months or
- Within 2 weeks of study vaccination for herbal products, vitamins, minerals, and over-the-counter medications.

Concomitant medications will be listed and summarized in a similar manner to that of prior medications.

For the purpose of inclusion in prior and concomitant medications tables, incomplete start and stop dates will be imputed according to the below rules (where UK, UKN, and UNKN indicate unknown or missing day, month, and year, respectively):

## **Missing Start Dates**

If day is missing and month and year are available:

• UK-MMM-YYYY: Assume 01-MMM-YYYY (first day of the month), but if month and year are the same as the first study vaccination month and year, then assume the date of first vaccination.

## If day and month are missing and year is available:

• UK-UKN-YYYY: Assume 01-JAN-YYYY (first day of the year), but if year is the same as the first study vaccination year, then assume the date of first study vaccination.

## If day, month and year (date) are missing:

UK-UKN-UNKN: Assume date of first study vaccination.

## **Missing Stop Dates**

If day missing and month and year are available:

• UK-MMM-YYYY: Assume the last day of the month

## If day and month are missing and year is available:

UK-UKN-YYYY: Assume 31-DEC-YYYY

#### If day, month and year (date) are missing:

• UK-UKN-UNKN: Do not impute and assume ongoing

(Note - In case of single dose vaccine or treatment, start date may be same as that of end date.)

#### 7.2. Study Treatments

#### 7.2.1. Extent of Exposure and Compliance

A listing of vaccine exposure will be provided to list participants. The listing will include assigned study vaccine, actual vaccine received, date and time of the vaccination and sorted by age group, dose group and participant number.

## 8. Analysis of Safety and Immunogenicity Study Objectives

## 8.1. Analysis of Primary Safety Objective

8.1.1. Analysis of solicited local and systemic AE up to 7 days after study vaccination (day 1-7), unsolicited AEs up to 28 days after study vaccination (day 1-28), abnormal clinical safety laboratory finding up to 8 days after study vaccination (day 1-8) and non-serious Covid-19 adverse events (Day 1 – study end)

The percentages of participants with at least one solicited local or systemic AE for 7 days following vaccination (day 1-7), participants with unsolicited AEs up to 28 days after study vaccination (day 1-28), participants with abnormal clinical safety laboratory findings up to 8 days after study vaccination (day 1-8) and non-serious Covid-19 adverse events (day 1 – study end) will be computed by dose group.

8.1.2. Analysis of Medically attended Adverse Events (MAAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) from study vaccination through the end of the study

Participants MAAEs and SAEs from study vaccination through the end of the study (approximately 180 days after the study vaccine administration, day 1-180) will be presented as the percentage of participants with such events throughout the study duration by dose and age group. Participants AESIs from study vaccination through the end of the study (day 1-180) will be presented by dose group.

## 8.2. Analysis of Secondary Immunogenicity Endpoints

8.2.1. GMTs of neutralizing Ab titer against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 and GMI from baseline of neutralizing Ab titers against pseudotyped bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection time point

For continuous variables and each dose group, summary statistics, geometric mean titer (GMT) and associated 95% CIs, and interquartile ranges will be provided. Listings will also be provided by age group, dose group, participant number and graphical presentations will be considered as needed.

Immunogenicity of the study vaccine will be assessed through GMTs at each collection time point (day 1) before the booster dose and after the booster dose (days 15, 29, 91, 181). GMTs and GMIs from baseline will be summarized with descriptive statistics including a bar chart (on log scale) for each age group versus time.

The GMT will be calculated using the following formula:

$$\left\{\frac{\sum_{i=1}^{n}\log_{10}(t_{i})}{n}\right\}$$

Where  $t_1, t_2, ..., t_n$  are n observed immunogenicity titers.

Statistical Analysis Plan Date Issued: 31JAN2023

The GMI measures the changes in immunogenicity titers or levels within participants (change from baseline in log titers). The GMI will be calculated using the following formula:

$$10^{\left\{\frac{\sum_{i=1}^{n}\log_{10}\left(v_{ij}/v_{ik}\right)}{n}\right\}} = 10^{\left\{\frac{\sum_{i=1}^{n}\log_{10}\left(v_{ij}\right) - \log_{10}\left(v_{ik}\right)}{n}\right\}}$$

where, for *n* participants,  $v_{ij}$  and  $v_{jk}$  are observed immunogenicity titers for participant *i* at time points *j* and *k*, k=baseline.

Antibody titers will be summarized at baseline and each postvaccination visit (the number of participants with nonmissing data, median, minimum, maximum, GMT, and 95% CI). Geometric mean increase and the corresponding 95% CI for the GMI as well as the minimum and maximum fold-rise value will be presented by age group or prior Covid-19 infection, dose group and visit. The 95% CI will be calculated based on the t-distribution of the log-transformed fold-rise values for GMTs and GMIs, then back-transformed to the original scale for presentation.

Supporting data listings will be provided for the All Enrolled Set by age group, dose group and participant number.

Bar charts (including 95% CIs) of GMT for serum IgG and NAb antibody levels by dose, age group, prior Covid-19 infection and visit will be provided in addition to summary tables.

The GMT at each postvaccination time point, the GMI from baseline, and the 95% CIs in all cohorts will be analyzed using an ANCOVA model on log10 transformed titers with dose group and age group as fixed in the model and prior Covid-19 infection and prevaccination baseline value as covariables.

8.2.2. Seroresponse rate 28 days after the booster dose (day 29), based on neutralizing Ab titers against pseudoviruses bearing S protein from SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants at each collection timepoint, with seroresponse defined as postboost titers ≥ 4× preboost titers.

Proportion of participants with neutralizing seroresponse of serum SARS-CoV-2 WT, Omicron BA.1, BA.2 and BA.5 variants specific Ab from baseline at day 29 by dose group and prior Covid-19 infection will be tabulated with 2-sided 95% Clopper Pearson CIs. The same summaries will be generated for seroresponse rate 14 days after booster dose (Day 15) as supportive analyses.









Statistical Analysis Plan Date Issued: 31JAN2023

## 9 Safety Analysis

Safety, tolerability, and reactogenicity will be assessed by clinical review of all relevant parameters including solicited and unsolicited AEs, SAEs, AESIs, MAAEs, AEs leading to withdrawal from study participation, safety laboratory test results, vital signs, and physical examination findings.

All safety analyses will be based on Safety Set. All safety analyses will be provided by dose group and age group unless otherwise specified.

#### 9.1 Adverse Events

An AE is any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to the IP. This definition includes exacerbations of pre-existing conditions. Stable pre-existing conditions which do not change in nature or severity during the study are not considered AEs; however, these should be reported as part of the medical history at screening.

SOC will be displayed in alphabetical order. PT will also be displayed alphabetically within SOC. Percentages will be based upon the number of participants in the Safety Set within each dose group.

Incomplete AE onset date/time and end date will be imputed following the rules below.

## **Missing Start Dates**

If day is missing and month and year are available:

• UK-MMM-YYYY: Assume 01-MMM-YYYY (first day of the month), but if month and year are the same as the first study vaccination month and year, then assume the date of first vaccination.

If day and month are missing and year is available:

• UK-UKN-YYYY: Assume 01-JAN-YYYY (first day of the year), but if year is the same as the first study vaccination year, then assume the date of first study vaccination.

#### If day, month and year (date) are missing:

UK-UKN-UNKN: Assume date of first study vaccination.

#### Missing Stop Dates

If day missing and month and year are available:

• UK-MMM-YYYY: Assume the last day of the month

If day and month are missing and year is available:

UK-UKN-YYYY: Assume 31-DEC-YYYY

If day, month and year (date) are missing:

UK-UKN-UNKN: Do not impute and assume ongoing

All adverse events will be classified by SOC and PT according to the MedDRA.

Statistical Analysis Plan Date Issued: 31JAN2023

Unless otherwise specified, AEs will be summarized by dose group based on Safety Set. A listing of AEs will be provided by age group, dose group and participant number.

All events from screening until vaccination will be considered as medical history.

## 9.1.1 Relationship of Adverse Events to Study Drug

Investigators will not be required to assess the causality of solicited AEs if the onset is during the solicitation period.

The investigator will determine the causal relationship between the study vaccine and the AE for all unsolicited AEs, SAE, MAAE and AESIs. The relationship of unsolicited AEs to the study vaccine (Yes, No) will be captured on the eCRF.

The number and percentage of participants along with the frequency of AEs (unsolicited AEs and SAEs) by SOC, PT, and relationship will be produced.

A participant with 2 or more AEs within the same SOC or PT level but different relationship will be counted only once in the level using the related incident. If the causality is missing, then a "missing" category will be included in the summary.

## 9.1.2 Severity of Adverse Event

The severity of AEs (mild, moderate, severe) will be captured on the eCRF. Adverse events (unsolicited AEs, solicited AEs, and SAEs) will be summarized including the number of participants and percentages by dose group, study vaccine, as well as by SOC, PT, and severity. If the severity is missing, then a "missing" severity category will be included in the summary. A participant with 2 or more AEs within the same SOC or PT level but different severity will be counted only once at the most severe level.

## 9.1.3 Outcome of Adverse Event

The outcome of an AE will be assessed as at the time of last observation per the following categories:

- Fatal
- Not Recovered/ Not Resolved
- Recovered/Resolved
- Recovered/Resolved with sequelae
- Recovering/Resolving
- Unknown

The number and percentage of participants along with the frequency of adverse events (unsolicited, AESIs, MAAEs and SAEs) will be summarized by SOC, PT, and outcome.

Statistical Analysis Plan Date Issued: 31JAN2023

A participant with 2 or more AEs within the same SOC or PT level but different outcome will be counted only once with higher outcome grading.

#### 9.1.4 Solicited Adverse Event

Solicited AEs are prespecified local and systemic. Solicited AEs will be collected from day 1 through 7 days following the vaccination (day 1-7) using eDiary. Solicited AEs with onset during the 7-day solicitation period that continue beyond the 7-day period will be reported as unsolicited AEs.

The following specific solicited adverse events will be used to assess reactogenicity.

Local reactions at injection site:

- Injection Site Pain
- Redness
- Swelling
- Lymphadenopathy (localized axillary, cervical or supraclavicular swelling or tenderness ipsilateral to the vaccination arm)

## Systemic reactions:

- Fever
- Headache
- Fatigue
- Myalgia
- Arthralgia
- Chills

The number and percentage of participants with any local solicited AEs, and systemic solicited AEs will be presented for each age group and dose group among participants with eDiary information available.

All solicited AEs local and systemic will be listed by age and participant number. Solicited adverse events reported until 7 days (day 1 through day 7) postvaccination will be summarized by maximum severity and by dose group.

Prolonged Solicited AEs that continue beyond day 7 will be reported on the eCRF as Unsolicited AEs and will be listed as such. The number and percentage of participants with prolonged solicited AE will be presented for each age group (any, any local, any systemic, each solicited AE).

In addition, the duration (in days) of solicited AEs which started within day 1-7 will be summarized by dose group for each age group. The duration for any severity will be calculated as Stop date – Start date + 1, where start date is the first day with AE while stop is the last day with the AE in or beyond the solicited period. The

Statistical Analysis Plan Date Issued: 31JAN2023

duration of solicited AE with specific severities (mild/moderate/severe, moderate/severe, severe) will be the number of days with the severity.

Currently on the eCRF the investigator can overwrite the severity of AEs on the eDiary, if he believes the event grading has not been recorded, has been underestimated or overestimated, and provide his assessment. When available the severity provided by the investigator will be used instead of the eDiary grading to generate the summaries of solicited events.

The percentage of eDiary days completed will be summarized by dose and age group. A day is considered completed in the eDiary if it was entered by the participant or the investigator. The percentage of completed days will be calculated as follows:

SumSymp/(7\*NumSymp\*ExpSubj)

SumSymp is the sum of the total number of days completed for a specific symptom across all symptoms and exposed subjects. NumSymp is the number of symptoms and ExpSubj is the number of exposed subjects.

#### 9.1.5 Unsolicited Adverse Event

Unsolicited AEs are defined as any AEs reported spontaneously by the participant, observed by the study staff during study visits or those identified during review of medical records or source documents. Solicited AEs with an onset after the 7-day solicitation period (day 1-7) will be considered unsolicited AEs. An unsolicited AE is defined as any AE that is volunteered from the participant and occurs within 28 days after vaccination (day 1-28).

The percentage of participants with unsolicited AEs onset date within day 1-28 will be provided by age group, dose group, by grade, outcome and causality (any, fatal, causally related, fatal/causally related).

The number and percentage of participants with unsolicited AEs onset date within day 1-28 will be provided by SOC and PT for each dose group (any grade, grade 3, related).

Unsolicited AEs will be summarized and listed up to day 28 after study vaccination (day 1-28).

A data listing for all Unsolicited AEs will be provided by age group, dose group and participant number.

#### 9.1.6 Adverse Events of Special Interest

An AESI (serious or nonserious) is defined as an AE or SAE of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor could be appropriate (ICH E2F; CIOMS VI).

Adverse events of special interest will include the following events:

Virologically confirmed Covid-19 (see protocol section 6.4 for definitions)

Statistical Analysis Plan Date Issued: 31JAN2023

- Potential immune-mediated disorders (see protocol section 13.4 for definitions)
- Anaphylaxis or severe hypersensitivity within 24 hours after study vaccine administration
- Myocarditis
- Pericarditis

AESIs will be identified using MedDRA queries and Investigator identification as per eCRF. Refer to appendix 15.3. MedDRA queries for identifying AESIs for details on these queries.

The percentage of participants with AESIs with onset date within day 1-28 and within day 1-180, identified by either the investigator or by MedDRA queries, will be provided by SOC and PT for each dose group.

Similarly, AESIs that are related to COVID-19 will be presented in a separate listing by age group, dose group and participant number.

AESIs will be reported until exit from study (up to day 180 after the study vaccine administration, day 1-180).

#### 9.1.7 Serious Adverse Events

An SAE is defined as any event that:

- Results in death
- Is immediately life-threatening
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect
- Is an important medical event that may not result in death, be life-threatening, or require hospitalization but, based upon appropriate medical judgment, jeopardizes the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse. All events of myocarditis and pericarditis will be considered important medical events and SAEs (see protocol section 6.1.3).

The percentage of participants with SAEs onset date within day 1-180 will be provided by dose group, by grade, outcome and causality.

The number and percentage of participants with SAE onset date within day 1-28 and within day 1-180 will be summarized by SOC, PT and casuality for each dose group (any, fatal, causally related, fatal/causally related).

SAEs will be summarized and listed from the time participant signs the ICF until exit from study (up to day 180 after the study vaccine administration, day 1-180).

A data listing for all SAEs will be provided by age group, dose group and participant number.

### 9.1.8 Medically Attended Adverse Events

Medically attended adverse events (MAAEs) is defined as an AE that results in a visit to a medical professional (eg, telephone call, physician's office visit, urgent care visit, emergency room visit or hospitalization). Scheduled study visits will not be considered medically attended visits. Medically attended adverse events related to study vaccination are to be reported from the time of first study vaccination until completion of the participant's last study-related procedure, which may include contact for safety follow-up.

The percentage of participants with MAAE onset date within day 1-180 will be provided by dose group and by grade.

All MAAEs and treatment-related MAAEs with onset date within day 1-28 and within day 1-180 will be presented in separate summary tables for each dose and age group and total by SOC and PT. All MAAEs will be presented in a data listing by age group, dose group and participant number.

MAAEs will be reported in both listings and summaries from the time participant signs the ICF until exit from study (up to day 180 after the study vaccine administration, day 1-180).

# **9.1.9 Adverse Events Leading to Treatment Discontinuation** Not applicable.

## 9.1.10 Adverse Events Leading to Study Discontinuation

Adverse events leading to study discontinuation are identified on the study disposition page of the eCRF by the AE number.

The number and percentage of participants with AE leading to discontinuation with onset date within day 1-28 will be summarized by SOC and PT for each dose group.

AEs leading to study discontinuation will be presented and a data listing will be provided by age group, dose group and participant number.

## 9.1.11 Death

The summary of AEs with an outcome of "Fatal" with onset date within day 1-180 will also be presented by SOC. The SOCs will presented alphabetically. Within each SOC, the PTs will be presented in alphabetical order.

All participants who have an AE with an outcome of "Death" will be presented in a listing by age group, dose group and participant number.

Deaths will be reported for both summaries and listings from the time participant signs the ICF until exit from study (up to day 180 after the study vaccine administration, day 1-180).

#### 9.2 Clinical Laboratory Evaluations

The following laboratory assessments will be performed:

| Hematology: | Basophils, eosinophils, erythrocytes (red blood cells), hemoglobin, |
|---|---|
| | leukocytes (white blood cells), lymphocytes, monocytes, neutrophils, |
| | and platelets |
| Chemistry: | Alanine aminotransferase, alkaline phosphatase, aspartate |
| | aminotransferase, total and direct bilirubin, blood urea nitrogen, and |
| | creatinine |
| SARS-CoV-2: | SARS-CoV-2 serology (antibody) will include N protein for |
| | prevaccination and postvaccination timepoints. |
| | SARS-CoV-2 RT-PCR (nasopharyngeal or mid-turbinate swab) |
| HIV/HBV/HCV | Hepatitis B surface antigen test |
| | HIV 4th generation antigen/Ab test |
| | Anti-HCV Ab test (and RNA test if anti-HCV Ab positive) |
| Other analyses: | Female participants of childbearing potential: |
| | <ul> <li>β-human chorionic gonadotropin (serum test at screening; urine</li> </ul> |
| | test at additional time points) |
| | Serum FSH, to confirm postmenopausal status |

Individual safety laboratory measurements for hematology, chemistry and coagulation laboratory panel will be provided. All listings will include the cohort, study vaccine, participants ID, laboratory test name result, date and time of measurements, reference range, and flag for measurements that are outside the reference range and sorted by age group, dose group and participant number.

Laboratory abnormalities will be graded for severity using the FDA toxicity grading table (DHHS 2007). Clinically relevant laboratory abnormalities will be reported as AEs using the AE grading.

A summary of patients with an abnormal laboratory value after study vacation (up to Day 8) will be presented. An abnormal laboratory is defined as any value outside of the normal range.

A by-participant listing will be provided for pregnancy test by age group, dose group and participant number.

## 9.3 Vital Sign Measurements

Vital sign measurements will include systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature. Observed values and changes from baseline will be summarized for each vital sign parameter by time point, and dose group.

Statistical Analysis Plan Date Issued: 31JAN2023

A supporting by-participant listing of vital sign parameters along with the investigator assessment will be provided by age group, dose group and participant number.

## 9.4 Physical Examination

A complete physical examination including height and weight will be performed at Screening. Symptomdirected physical examinations will be performed as clinically indicated at subsequent visits. The results of the physical examination findings will be listed by participants and dose group, and sorted by age group, dose group and participant number.

## 9.5 Electrocardiogram

At screening and at the Day 8 visit, all participants will be assessed by 12-lead ECG for evidence of asymptomatic myocarditis or pericarditis. The results of the electrocardiogram findings will be listed by participants and dose group, and sorted by age group, dose group and participant number.

#### 10 Pharmacokinetics

Not applicable.

## 11 Pharmacodynamics

Not applicable.

## 12 Interim Analysis

There are 2 planned interim analyses of safety and immunogenicity data for at least neutralizing Ab titers against SARS-CoV-2 WT, Omicron BA.1 or BA.5 variant pseudoviruses. A first interim analysis of safety and immunogenicity data covering at least neutralizing Ab titers against pseudovirus bearing S protein from WT, Omicron BA.1 or BA.5 SARS-CoV-2 up to 14 days after study vaccine administration in participants enrolled in Cohorts 1, 2, and 3 will be performed including at least day 1 and day 15 data. A second interim analysis of safety and immunogenicity data covering at least neutralizing Ab titers against pseudovirus bearing S protein from WT, Omicron BA.1, or BA.5 SARS-CoV-2 will be performed 14 days after participants in Cohorts 4 and 5 have received study vaccine including at least day 1 and day 15 data in Cohorts 4 and 5 and day 29 data in addition in Cohorts 1,2 and 3.

Further to the above the first interim will be based on the PNA data. Available binding IgG data at the time of the first interim will be included, but it is not requested to have 100% of these data at the time of the first interim analysis. For PNA, BA.1, BA.5 and Wuhan (ancestral strain, comparator with CV2CoV) will be prioritized (priority #1). BA.2 can be done as priority #2. Regarding cohort 6 and 7 (lowest doses), it is unsure at this stage whether these cohorts will be enrolled as it will depend on the data generated at 12 mcg.

The safety set will be used for the interim immunogenicity analyses.

Statistical Analysis Plan Date Issued: 31JAN2023

## 13 Changes in the Planned Analysis

Because the assays are not fully validated values below LLOQ or above ULOQ they will be used as released. Results released as below a value will be assigned 0.5\*the value. Results released as above a value will be assigned the value.

## 14 References

Department of Health and Human Services (DHHS), Food and Drug Administration, Center for Biologics Evaluation and Research (US). Guidance for industry. Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine clinical trials. September 2007 [cited 2021 Jul 09]. Available from: <a href="https://www.fda.gov/media/73679/download">https://www.fda.gov/media/73679/download</a>

World Health Organization (WHO). WHO coronavirus (COVID-19) dashboard [Internet]. 2021 [cited 2021 Jul 07]. Available from: <a href="https://covid19.who.int/">https://covid19.who.int/</a>

Statistical Analysis Plan Date Issued: 31JAN2023

# 15 Appendices

## 15.1 Schedule of Events

| | Screeninga | D1 | D4 | D8 | D15 | D29 | D91 | D181<br>(EOS) | ET<br>Visit | Unscheduled<br>Visit for<br>Suspected<br>COVID19 | Unscheduled<br>COVID-19<br>Convalescent<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Window | D-14 to -1 | 0 | ±1 | ±1 | ±3 | ±3 | ±5 | ±7 | NA | NA | NA |
| Visit | 1 | 2 | Phone | 3 | 4 | 5 | 6 | 7 | NA | NA | NA |
| Informed consent | X | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | |
| Reassess study vaccine eligibility <sup>b</sup> | | X | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history (including vaccination history) | X | | | | 1 | | , | | | | |
| Pregnancy test <sup>c</sup> | X | X | | | | | | | | | |
| CCI | | | | | | | | | | | |
| Physical examination <sup>f</sup> | X | X | | X | X | X | X | X | X | X | X |
| Vital sign measurements <sup>g</sup> | X | X | | X | X | X | X | X | X | X | X |
| Viral screening assaysh | X | | | | | | | | | | |
| Hematology and serum chemistryh | X | $X^d$ | | X | | | | | | | |
| CCI | | | | | | | | | | | |
| Group assignment for Part A/<br>Randomization for Part B | | X | | | | | | | | | |
| Initiate eDiary for solicited AEs <sup>i</sup> | | X | | | | | | | | | |
| 12-lead ECG examination | X | | | X | | | | | | | |
| Site staff review of eDiary | | | X | X | | | | | | | |
| CCI | | | | | | | | | | | |
| COVID-19 assessment <sup>k</sup> | | | | | | | | | | $X^k$ | X <sup>k</sup> |

#### 31 Jan 2023 Statistical Analysis Plan 3 | VV-TMF-8850143 | 1.0

GlaxoSmithKline Biologicals SA CV2 SARS-CV0501-012 BST (218595) Statistical Analysis Plan Date Issued: 31JAN2023

Note: Due to the ongoing pandemic, follow-up visits may be completed via telephone calls, consistent with local regulations.

- a. If the investigator believes there is a reasonable justification to do so, all screening procedures may be repeated (maximum 1 rescreening per participant is allowed). Only results from the rescreening visit, if it occurs, will be taken into consideration and recorded in the eCRF. The participant can only be vaccinated once the investigator receives the results and confirms the eligibility criteria.
- b. Prior to study vaccine administration, participants will be reassessed for development of any new condition that would be considered exclusionary including acute illness or pregnancy. Assessment will be based on pregnancy test results, participant-reported symptomology, vital sign measurements, and physical examination findings.
- c. A serum pregnancy test will be performed at screening in WOCBP. A urine pregnancy test by dipstick will be performed prior to study vaccination. Negative confirmation is required prior to study vaccine administration. Pregnancy test may be repeated at an unscheduled visit per investigator's discretion.
- d. On day 1, the blood sample should be collected *before* study vaccine administration.
- e. CC
- f. A complete physical examination including height and weight will be performed at screening. Symptom-directed physical examinations will be performed as clinically indicated at subsequent visits.
- g. Vital sign measurements (temperature, pulse rate, oxygen saturation by pulse oximetry, respiration rate, and blood pressure) should be collected before and after study vaccination on D1. Vital sign measurements should be performed before any scheduled blood collection. Participants who are febrile (temperature ≥38.0°C or ≥100.4°F) before study vaccination on D1 should be rescheduled for study vaccination within the relevant window period.
- h. Clinical safety laboratory testing will include hematology and serum chemistry. Screening laboratory tests may be repeated once for enrollment requirements. At unscheduled visits, clinical safety laboratory testing may be performed per investigator's discretion. Viral screening assays include HIV1/2 Antigen/Ab, hepatitis B surface antigen (HBsAg) and hepatitis C virus antibodies (HCV Abs). Testing for HCV RNA will be performed in participants who test positive for HCV Ab.
- i. An eDiary will be initiated for daily recording by the participant of solicited local and systemic adverse events.
- j. Solicited local and systemic AEs will be collected during the 7 days after study vaccination via eDiaries. Unsolicited AEs will be collected for 28 days after study vaccination. SAEs, MAAEs, and AESIs will be collected for the duration of the study.
- k. All suspected cases of COVID-19 in study participants will be diagnosed and clinically evaluated according to the definitions provided in Section 6.1.2. Such participants may have unscheduled study site visits and nasopharyngeal RT-PCR testing for SARS-CoV-2. An unscheduled visit may be performed for participants reporting symptoms consistent with COVID-19. An initial visit should be scheduled upon report of symptom onset, preferably within 3 days of symptom onset. Alternatively, an investigator may utilize participant medical records from non-study care providers to verify whether a participant was infected with SARS-CoV-2. An additional unscheduled, COVID-19 convalescent visit will be preferably conducted within the month after the participant is confirmed with COVID-19. At the convalescent visit, the investigator will seek medical records documenting any treatments and hospitalizations related to COVID-19.



# 15.3. MedDRA queries for identifying AESIs

The tables below are MedDRA version specific and may be revised with a new MedDRA version:

Table 15 1 Preferred terms for AESIs which are not pIMDs

| | Autoimmune myocarditis |
|---|---|
| | Eosinophilic myocarditis |
| Myggarditis | Giant cell myocarditis; |
| Myocarditis | Hypersensitivity myocarditis |
| | Immune-mediated myocarditis |
| | Myocarditis |
| | Autoimmune pericarditis |
| | Pericarditis |
| Pericarditis | Pericarditis adhesive |
| | Pericarditis constrictive |
| | Pleuropericarditis |
| Severe Hypersensitivity | Grade 3 unsolicited AEs under MedDRA SMQ |
| | hypersensitivity, narrow search (includes anaphylaxis), with an |
| | onset within 24 hours after vaccination |

COVID 19 infection will be based on PCR test (there is no MEDRA query)

Table 15 2 Preferred terms for AESIs which are pIMDs

| Event Category | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| Neuroinflammatory | Cranial nerve disorders | Anosmia | 10002653 |
| disorders | and inflammations | IIIrd nerve paralysis | 10021283 |
| | | IIIrd nerve paresis | 10054202 |
| | | IVth nerve paralysis | 10023110 |
| | | IVth nerve paresis | 10054201 |
| | | Trigeminal palsy | 10049788 |
| | | Trigeminal nerve paresis | 10068008 |
| | | VIth nerve paralysis | 10047641 |
| | | VIth nerve paresis | 10071044 |
| | | Facial paralysis | 10016062 |
| | | Facial paresis | 10051267 |
| | | Acoustic neuritis | 10063162 |
| | | Glossopharyngeal nerve paralysis | 10051270 |
| | | Tongue paralysis | 10043972 |
| | | Vagus nerve paralysis | 10064661 |
| | | Vocal cord paralysis | 10047674 |
| | | Vocal cord paresis | 10049234 |
| | | XIth nerve paralysis | 10048842 |
| | | Hypoglossal nerve paralysis | 10069450 |
| | | Hypoglossal nerve paresis | 10067129 |
| | | Bulbar palsy | 10006542 |
| | | Oculofacial paralysis | 10030069 |
| | | Neuritis cranial | 10029244 |
| | | Cranial nerve disorder | 10061093 |
| | | Paresis cranial nerve | 10061911 |
| | A | Cranial nerve paralysis | 10061908 |
| | | Cranial nerve palsies multiple | 10011314 |
| | | Optic neuritis | 10030942 |
| | Multiple sclerosis | Multiple sclerosis | 10028245 |
| | Triangle strategie | Radiologically isolated syndrome | 10079292 |
| | | Primary progressive multiple sclerosis | 10063401 |
| | | Progressive multiple sclerosis | 10053395 |
| | <b>y</b> | Marburg's variant multiple sclerosis | 10067067 |
| | | Secondary progressive multiple sclerosis | 10063400 |
| | | Multiple sclerosis relapse | 10048393 |
| | | Relapsing multiple sclerosis | 10080700 |
| | | Multiple sclerosis relapse prophylaxis | 10070495 |
| | | Progressive relapsing multiple sclerosis | 10067063 |
| | | Relapsing-remitting multiple sclerosis | 10063399 |
| | | Tumefactive multiple sclerosis | 10078556 |
| | | Expanded disability status scale score decreased | 10071385 |
| | | Expanded disability status scale score increased | 10071384 |
| | Myelitis / Transverse | Myelitis transverse | 10071384 |
| | myelitis | Myelitis | 10028524 |
| | injoinis | Acute flaccid myelitis | 10028324 |
| | | Noninfectious myelitis | 10082097 |
| | Guillain Darrá armárama | | |
| | Guillain-Barré syndrome | Guillain-Barré syndrome | 10018767 |
| | A auto disconsinate 1 | Miller Fisher syndrome | 10049567 |
| | Acute disseminated | Demyelination Learners 1 and 1 | 10012305 |
| | encephalomyelitis and | Intramyelinic oedema | 10083038 |

| <b>Event Category</b> | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| | demyelination (including | Autoimmune demyelinating disease | 10075688 |
| | site specific variants) | Clinically isolated syndrome | 10071068 |
| | | Leukoencephalomyelitis | 10048999 |
| | | Leukoencephalopathy | 10024382 |
| | | Acute disseminated encephalomyelitis | 10000709 |
| | | Acute haemorrhagic leukoencephalitis | 10058994 |
| | | Concentric sclerosis | 10010252 |
| | | Encephalitis periaxialis diffusa | 10049020 |
| | | Limbic encephalitis | 10078012 |
| | | Neuromyelitis optica spectrum disorder | 10077875 |
| | | Neuromyelitis optica pseudo relapse | 10080353 |
| | | Autoimmune encephalopathy | 10075691 |
| | | Bickerstaff's encephalitis | 10076985 |
| | | Noninfective encephalitis | 10074712 |
| | | Encephalitis autoimmune | 10072378 |
| | | Immune-mediated encephalitis | 10083074 |
| | | Rasmussen encephalitis | 10071141 |
| | | Encephalitis allergic | 10056387 |
| | | Encephalitis brain stem | 10048997 |
| | | Encephalitis haemorrhagic | 10014589 |
| | | Encephalomyelitis | 10014619 |
| | | Noninfective encephalomyelitis | 10074713 |
| | | Encephalitis post immunisation | 10014602 |
| | | Panencephalitis | 10056332 |
| | | Encephalitis toxic | 10014607 |
| | | Chronic lymphocytic inflammation with pontine perivascular enhancement responsive to steroids | 10075197 |
| | Myasthenia gravis | Myasthenia gravis | 10028417 |
| | | Myasthenia gravis crisis | 10062758 |
| | | Ocular myasthenia | 10049168 |
| | | Myasthenic Syndrome | 10028424 |
| | Autoimmune / Immune- | Autoimmune neuropathy | 10070439 |
| | mediated peripheral | Immune-mediated neuropathy | 10078963 |
| | neuropathies and | Neuritis | 10029240 |
| | plexopathies | Anti-myelin-associated glycoprotein associated polyneuropathy | 10078324 |
| | | Subacute inflammatory demyelinating polyneuropathy | 10081726 |
| | | Chronic inflammatory demyelinating polyradiculoneuropathy | 10057645 |
| | | Lewis-Sumner syndrome | 10065580 |
| | | Demyelinating polyneuropathy | 10061811 |
| | | Polyneuropathy idiopathic progressive | 10036111 |
| | | Multifocal motor neuropathy | 10055111 |
| | | Acute motor-sensory axonal neuropathy | 10003373 |
| | | Acute motor axonal neuropathy | 10076658 |
| | | Cervical neuritis | 10070038 |
| | | Mononeuritis | 10003293 |
| | | Mononeuropathy multiplex | 10027918 |
| | | Brachial plexopathy | 10027918 |
| | | Radiculitis brachial | 10003417 |
| | | Neuralgic amyotrophy | 10037778 |
| | Narcoloney | | 10029229 |
| | Narcolepsy | Narcolepsy | 10028/13 |

| Event Category | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| Musculoskeletal | Systemic lupus | Systemic lupus erythematosus | 10042945 |
| disorders | erythematosus | SLE arthritis | 10040968 |
| | | Cutaneous lupus erythematosus | 10056509 |
| | | Acute cutaneous lupus erythematosus | 10057928 |
| | | Chronic cutaneous lupus erythematosus | 10057929 |
| | | Subacute cutaneous lupus erythematosus | 10057903 |
| | | Lupus cystitis | 10074714 |
| | | Lupus encephalitis | 10025130 |
| | | Lupus endocarditis | 10058225 |
| | | Lupus enteritis | 10067738 |
| | | Lupus hepatitis | 10067737 |
| | | Lupus myocarditis | 10066391 |
| | | Lupus myositis | 10079642 |
| | | Lupus nephritis | 10025140 |
| | | Lupus pancreatitis | 10067750 |
| | | Lupus pleurisy | 10073694 |
| | | Lupus pneumonitis | 10057481 |
| | | Lupus-like syndrome | 10050551 |
| | | Neuropsychiatric lupus | 10063663 |
| | | Central nervous system lupus | 10076328 |
| | | Pericarditis lupus | 10058149 |
| | | Peritonitis lupus | 10062898 |
| | | Systemic lupus erythematosus rash | 10042946 |
| | | Systemic lupus erythematosus disease activity index abnormal | 10067659 |
| | 1 | Systemic lupus erythematosus disease activity index decreased | 10067658 |
| | | Systemic lupus erythematosus disease activity index increased | 10067657 |
| | Systemic Scleroderma | Scleroderma | 10039710 |
| | (Systemic sclerosis) | Scleroderma renal crisis | 10062553 |
| | | Scleroderma associated digital ulcer | 10073229 |
| | V 7 | Reynold's syndrome | 10070953 |
| | | Systemic sclerosis pulmonary | 10042954 |
| | Y | Systemic scleroderma | 10078638 |
| | | Anti-RNA polymerase III antibody increased | 10082280 |
| | | Anti-RNA polymerase III antibody positive | 10082283 |
| | | CREST syndrome | 10011380 |
| | Muscular Autoimmune / | Polymyalgia rheumatica | 10036099 |
| | Immune-mediated | Dermatomyositis | 10030033 |
| | disorders | Polymyositis | 10036102 |
| | | Autoimmune myositis | 10030102 |
| | | Immune-mediated myositis | 10083073 |
| | | Juvenile polymyositis | 10083073 |
| | | Antisynthetase syndrome | 100/00/3 |
| | Rheumatoid arthritis and | Rheumatoid arthritis | 10039073 |
| | associated conditions | Autoimmune arthritis | 10039073 |
| | associated conditions | Immune-mediated arthritis | 10071133 |
| | | Laryngeal rheumatoid arthritis | 10083133 |
| | | Rheumatoid lung | _ |
| | | Rheumatoid scleritis | 10039081<br>10067427 |
| | | Rheumatic brain disease | |
| | | Aneumane oram disease | 10079411 |

| <b>Event Category</b> | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| | | Rheumatoid neutrophilic dermatosis | 10072362 |
| | | Rheumatoid nodule | 10048694 |
| | | Juvenile idiopathic arthritis | 10059176 |
| | | Cogan's syndrome | 10056667 |
| | | Palindromic rheumatism | 10033534 |
| | | Still's disease | 10042061 |
| | Spondyloarthropathies | Arthritis reactive | 10003267 |
| | | Reiter's syndrome | 10038294 |
| | | Ankylosing spondylitis | 10002556 |
| | | Spondylitis | 10061371 |
| | | Spondyloarthropathy | 10051265 |
| | | Juvenile spondyloarthritis | 10076675 |
| | | Enteropathic spondylitis | 10076549 |
| | | Psoriatic arthropathy | 10037162 |
| | | Juvenile psoriatic arthritis | 10076674 |
| | Relapsing polychondritis | Polychondritis | 10065159 |
| | Mixed connective tissue | Overlap syndrome | 10068786 |
| | disease | Mixed connective tissue disease | 10027754 |
| | Gout | Gout | 10018627 |
| | | Gouty arthritis | 10018634 |
| | | Gouty tophus | 10018641 |
| Gastrointestinal | Inflammatory Bowel | Crohn's disease | 10011401 |
| disorders | disease | Colitis ulcerative | 10009900 |
| | | Colitis microscopic | 10056979 |
| | | Autoimmune colitis | 10075761 |
| | | Immune-mediated enterocolitis | 10078961 |
| | | Inflammatory bowel disease | 10021972 |
| | | Arthritis enteropathic | 10003253 |
| | | Proctitis ulcerative | 10036783 |
| | | Autoimmune enteropathy | 10081456 |
| | Autoimmune / Immune- | Autoimmune pancreatitis | 10069002 |
| | mediated pancreatitis | Immune-mediated pancreatitis | 10083072 |
| | Celiac disease | Coeliac disease | 10009839 |
| Liver disorders | Autoimmune / Immune- | Autoimmune hepatitis | 10003827 |
| | mediated hepatobiliary | Immune-mediated hepatitis | 10078962 |
| | diseases | Biliary cirrhosis primary | 10004661 |
| | | Primary biliary cholangitis | 10080429 |
| | | Cholangitis sclerosing | 10008609 |
| Endocrine and | Autoimmune / immune- | Autoimmune hypothyroidism | 10076644 |
| Metabolic disorders | mediated thyroid diseases | Immune-mediated hypothyroidism | 10083075 |
| | | Atrophic thyroiditis | 10077172 |
| | | Autoimmune thyroiditis | 10049046 |
| | | Immune-mediated thyroiditis | 10083071 |
| | | Silent thyroiditis | 10079012 |
| | | Hashimoto's encephalopathy | 10069432 |
| | | Hashitoxicosis | 10067873 |
| | | Basedow's disease | 10004161 |
| | | Marine Lenhart syndrome | 10068828 |
| | | Autoimmune thyroid disorder | 10079165 |
| | Autoimmune / Immune- | Autoimmune endocrine disorder | 10078953 |
| | mediated endocrinopathy | Immune-mediated endocrinopathy | 10078964 |
| | (NOS) | | |

| <b>Event Category</b> | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| | Diabetes mellitus type I | Type 1 diabetes mellitus | 10067584 |
| | | Fulminant type 1 diabetes mellitus | 10072628 |
| | Polyglandular autoimmune | Polyglandular autoimmune syndrome type I | 10036072 |
| | syndrome | Polyglandular autoimmune syndrome type II | 10036073 |
| | | Polyglandular autoimmune syndrome type III | 10064115 |
| | Autoimmune hypophysitis | Lymphocytic hypophysitis | 10063685 |
| | Addison's disease | Addison's disease | 10001130 |
| Skin disorders | Psoriasis | Psoriasis | 10037153 |
| | Vitiligo | Vitiligo | 10047642 |
| | Erythema nodosum | Erythema nodosum | 10015226 |
| | Alopecia areata | Alopecia areata | 10001761 |
| | Lichen planus | Lichen planopilaris | 10081142 |
| | | Lichen planus | 10024429 |
| | Sweet's syndrome | Acute febrile neutrophilic dermatosis | 10000748 |
| | Autoimmune / Immune- | Pemphigus | 10034280 |
| | mediated bullous skin | Pemphigoid | 10034277 |
| | diseases | Dermatitis herpetiformis | 10012468 |
| | | Autoimmune dermatitis | 10075689 |
| | | Immune-mediated dermatitis | 10083156 |
| | Localised Scleroderma | Morphoea | 10027982 |
| Vasculitides | Vasculitis and vasculitides | Acute haemorrhagic oedema of infancy | 10070599 |
| | | Administration site vasculitis | 10075969 |
| | | Anti-neutrophil cytoplasmic antibody positive vasculitis | 10050894 |
| | Ó | Aortitis | 10002921 |
| | | Application site vasculitis | 10076027 |
| | | Arteritis | 10003230 |
| | | Arteritis coronary | 10003232 |
| | | Behcet's syndrome | 10004213 |
| | | Capillaritis | 10068406 |
| | | Central nervous system vasculitis | 10081778 |
| | | Cerebral arteritis | 10008087 |
| | | Chronic pigmented purpura | 10072726 |
| | | Cutaneous vasculitis | 10011686 |
| | | Diffuse vasculitis | 10012978 |
| | , | Eosinophilic granulomatosis with polyangiitis | 10078117 |
| | | Erythema induratum | 10015213 |
| | | Granulomatosis with polyangiitis | 10072579 |
| | | Haemorrhagic vasculitis | 10071252 |
| | | Henoch-Schonlein purpura | 10019617 |
| | | Henoch-Schonlein purpura nephritis | 10069440 |
| | | Hypersensitivity vasculitis | 10020764 |
| | | Injection site vasculitis | 10067995 |
| | | Kawasaki's disease | 10023320 |
| | | Langerhans' cell histiocytosis | 10023320 |
| | | Lupus vasculitis | 10058143 |
| | | MAGIC syndrome | 10078132 |
| | | Microscopic polyangiitis | 100/3132 |
| | | Nodular vasculitis | 10003344 |
| | | Ocular vasculitis | 10029491 |
| | | Optic ischaemic neuropathy | 10030924 |
| | | Optic neuropathy | 10030924 |
| | | Polyarteritis nodosa | |
| | | rotyatienus nodosa | 10036024 |

| Event Category | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| | | Pulmonary vasculitis | 10037457 |
| | | Renal arteritis | 10038373 |
| | | Renal vasculitis | 10038546 |
| | | Retinal vasculitis | 10038905 |
| | | Rheumatoid vasculitis | 10048628 |
| | | Segmented hyalinising vasculitis | 10067527 |
| | | Takayasu's arteritis | 10043097 |
| | | Temporal arteritis | 10043207 |
| | | Thromboangiitis obliterans | 10043540 |
| | | Urticarial vasculitis | 10048820 |
| | | Vaccination site vasculitis | 10076191 |
| | | Vascular purpura | 10047097 |
| | | Vasculitic rash | 10047111 |
| | | Vasculitic ulcer | 10075714 |
| | | Vasculitis | 10047115 |
| | | Vasculitis gastrointestinal | 10048319 |
| | | Vasculitis necrotising | 10047124 |
| Other | Stevens-Johnson syndrome | Stevens-Johnson syndrome | 10042033 |
| | | Erythema multiforme | 10015218 |
| | | Toxic epidermal necrolysis | 10044223 |
| | | SJS-TEN overlap | 10083164 |
| | Blood autoimmune / | Autoimmune anaemia | 10080243 |
| | immune-mediated disoders | Autoimmune haemolytic anaemia | 10073785 |
| | | Warm type haemolytic anaemia | 10047822 |
| | | Cold type haemolytic anaemia | 10009868 |
| | | Coombs positive haemolytic anaemia | 10010941 |
| | | Evans syndrome | 10053873 |
| | | Immune thrombocytopenic purpura | 10074667 |
| | | Thrombocytopenic purpura | 10043561 |
| | | Thrombotic thrombocytopenic purpura | 10043648 |
| | | Autoimmune aplastic anaemia | 10071576 |
| | | Autoimmune neutropenia | 10055128 |
| | Y ' | Autoimmune pancytopenia | 10069509 |
| | | Immune-mediated pancytopenia | 10083004 |
| | The state of the s | Antiphospholipid syndrome | 10002817 |
| | | Pernicious anaemia | 10034695 |
| | Autoimmune / immune- | Glomerulonephritis rapidly progressive | 10018378 |
| | mediated | IgA nephropathy | 10021263 |
| | glomerulonephritis | IgM nephropathy | 10077209 |
| | | C1q nephropathy | 10081461 |
| | | Glomerulonephritis membranous | 10018372 |
| | | Glomerulonephritis membranoproliferative | 10018370 |
| | | Membranous-like glomerulopathy with masked IgG- | 10083098 |
| | | kappa deposits | 100000 |
| | | Mesangioproliferative glomerulonephritis | 10066453 |
| | | Anti-glomerular basement membrane disease | 10081981 |
| | | Autoimmune nephritis | 10077087 |
| | | Immune-mediated nephritis | 10083070 |
| | | Chronic autoimmune glomerulonephritis | 10073016 |
| | | Tubulointerstitial nephritis and uveitis syndrome | 10069034 |
| | Ocular autoimmune / | Uveitis | 10046851 |
| | immune-mediated diseases | Vogt-Koyanagi-Harada disease | 10082001 |

| Event Category | Immune-Mediated<br>Disorder | MedDRA PT | PT Code |
|---|---|---|---|
| | | Ocular pemphigoid | 10067776 |
| | | Autoimmune retinopathy | 10071578 |
| | | Acute macular outer retinopathy | 10079367 |
| | | Autoimmune uveitis | 10075690 |
| | | Immune-mediated uveitis | 10083069 |
| | | Autoimmune eye disorder | 10081123 |
| | Autoimmune / immune- | Autoimmune myocarditis | 10064539 |
| | mediated heart disease | Immune-mediated myocarditis | 10082606 |
| | | Autoimmune pericarditis | 10079058 |
| | Sarcoidosis | Sarcoidosis | 10039486 |
| | | Pulmonary sarcoidosis | 10037430 |
| | | Neurosarcoidosis | 10078011 |
| | | Cutaneous sarcoidosis | 10011674 |
| | | Liver sarcoidosis | 10068664 |
| | | Muscular sarcoidosis | 10028365 |
| | | Ocular sarcoidosis | 10065700 |
| | Sjögren's syndrome | Sjogren's syndrome | 10040767 |
| | Autoimmune lung disease | Idiopathic pulmonary fibrosis | 10021240 |
| | | Idiopathic interstitial pneumonia | 10078268 |
| | | Interstitial lung disease | 10022611 |
| | | Pulmonary fibrosis | 10037383 |
| | | Autoimmune lung disease | 10080701 |
| | | Immune-mediated pneumonitis | 10082452 |
| | Goodpasture's syndrome | Goodpasture's syndrome | 10018620 |
| | Raynaud's phenomenon | Raynaud's phenomenon | 10037912 |